CLINICAL TRIAL: NCT05483894
Title: Atorvastatin Use and Portal Hypertension in Patients With Hepatitis B Virus-related Liver Cirrhosis: A Randomized Controlled Trial
Acronym: STAPH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Dong Hyun Sinn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC 2021-06-205-001
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B; Portal Hypertension
Keywords: Atorvastatin; HBV- Related Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Hepatitis B; Hypertension, Portal | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Atorvastatin 10mg once daily for 24 weeks
  Interventions: Drug: Atorvastatin 10mg
- Control group (Placebo Comparator): Placebo once daily for 12 weeks and then Atorvastatin 10mg once daily for 12 weeks
  Interventions: Drug: Atorvastatin 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin 10mg(Lipinon Tab. 10mg) once daily for 24 weeks for experimental group
  Other Names: Lipinon Tab. 10mg
Drug: Placebo — Placebo once daily for 12 weeks and than Atorvastatin(Lipinon Tab. 10mg) for 12 weeks for control group
  Arms: Control group

SUMMARY:
To evaluate whether atorvastatin can improve portal hypertension in patients with chronic hepatitis B related compensated cirrhosis with portal hypertension

DETAILED DESCRIPTION:
In order to derive a reliable correlation between statin use and the reduction of portal hypertension, it is necessary to proceed with a clinical study with a high level of evidence, such as a randomized controlled clinical trial study. In addition, previous small randomized controlled trials had a limitation in that patients with various causes of liver cirrhosis were included. In this study, only patients diagnosed with chronic hepatitis B and compensated cirrhosis who are taking antiviral treatment will be included in the study, and in patients whose viral activity are suppressed by taking antiviral treatment, it was investigated whether statin administration had a significant effect in additionally improving portal pressure. We want to prove it through a randomized controlled clinical trial study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 19 and 69 years of age
2. If HBsAg positivity has been observed for more than 6 months or a clinical history of chronic hepatitis B is confirmed
3. When liver cirrhosis is diagnosed histologically, radiologically, or clinically (if one or more of A-D is applicable) A. When stage F4 fibrosis is confirmed by liver biopsy B. When splenomegaly is observed with morphological changes (surface nodularity and hypertrophy of the caudate lobe) appropriate for liver cirrhosis.

   C. If the platelet count is less than 100,000/mm3 in two consecutive tests D. When esophageal varices or gastric varices are confirmed by upper gastrointestinal endoscopy
4. If the serum HBV DNA is well controlled to 2000 International Unit (IU)/mL or less while taking antiviral treatment
5. When the splenic elasticity measured by two-dimensional shear wave elastography is greater than 25 kilopascal(kPa)
6. When informed consent is possible

Exclusion Criteria:

1. Hepatitis C or HIV co-infected person
2. Those who continuously drink more than the standard (alcohol intake exceeding 20g per day)
3. In case of decreased liver function with Child Pugh score of 7 or higher
4. History of decompensated cirrhosis: history of ascites, spontaneous bacterial peritonitis, hepatic coma, varicose bleeding, hepatic nephrotic syndrome
5. If there is a history of cancer (except for cases where there is no recurrence for 5 years after treatment due to early solid organ tumors (early gastric cancer, thyroid cancer))
6. If there is a serious comorbidity whose life expectancy is estimated to be less than 3 years
7. In case of chronic kidney disease estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2
8. If portal vein thrombosis is diagnosed
9. Previous intrahepatic portal vein shunt intervention or liver transplantation
10. A history of statin administration within the last 2 years
11. In case of side effects from previous statin administration (drug-related hepatotoxicity, muscle toxicity, allergic reaction, etc.)

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Response rate of 12 weeks of atorvastatin in experimental group and 12 weeks of placebo in control group | 12 weeks
  A responder is defined as a case in which the percentage change in spleen stiffness decreased by 10% or more from baseline after 12 weeks of atorvastatin or placebo administration. When the ratio of the number of responders to the number of participants in each group is defined as the response rate, there is a difference in the response rates between the experimental group and the control group.

SECONDARY OUTCOMES:
Response rate of 12 weeks of atorvastatin in experimental group and 24 weeks of atorvastatin in experimental group | 24 weeks
  After 12 weeks of atorvastatin administration, the response rate of the experimental group in which the percentage change in spleen stiffness decreased by 10% or more compared to the baseline value after 12 weeks of administration is different from the response rate after 24 weeks of the experimental group, in which the percentage change in spleen stiffness decreased by more than 10% compared to the baseline after 24 weeks of administration.
Response rate of 12 weeks of placebo in control group and 24 weeks of atorvastatin in experimental group | 24 weeks
  The response rate after 12 weeks of placebo administration in the control group is different from the response rate after 24 weeks of atorvastatin administration in the experimental group.
Response rate of 12 weeks of placebo in control group and 12 weeks of atorvastatin in control group | 12 weeks
  The response rate after 12 weeks of placebo administration in the control group is different from the response rate after 12 weeks of atorvastatin administration (24 weeks after the start of the study) in the control group at 12 weeks.
Adverse events | 24 weeks
  Frequency of adverse events (hepatotoxicity, muscle toxicity) after atorvastatin administration